CLINICAL TRIAL: NCT04741321
Title: Cross-cultural Adaptation and Validation of the VascuQol-6 Spanish Version
Brief Title: Validation of VascuQol-6 Spanish Version
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: VALVAS
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-test group: After translation to Spanish, VQ-6 questionnaire is given to 20 patients to assess understanding by the patient.
  Interventions: Other: VascuQol-6 questionnaire Spanish version
- Test and re-test group: 80 patients will be recruited to answer VQ-6 questionnaire and SF-12 questionnaire. After 3-4 weeks, these patients will be re-asked with the same questionnaires.
  Interventions: Other: VascuQol-6 questionnaire Spanish version

INTERVENTIONS:
Other: VascuQol-6 questionnaire Spanish version — VascuQol-6 questionnaire was translated by two professional translators into Spanish.

SUMMARY:
VascuQol (VQ) is a specific questionnaire to assess the quality of life of patients with critical limb ischemia which is also used as an index in vascular registries. The original version has 25 items (VQ-25), divided into 5 subscales or domains: pain, symptoms, activity, social and emotional. The shortened version, VascuQol-6 (VQ-6) is made up of 6 questions and 4 possible answers, which score from 1 (worst quality of life perceived by the patient) to 4 (best quality of life perceived by the patient). The total score is between 6 and 24, and a higher value is related to better health.

While the VQ-25 questionnaire has been translated and validated in 21 languages, the shortened version VQ-6 has been translated and validated in some languages, not including Spanish. As it is a fast and easy-to-use tool iwhich has demonstrated statistical validation to measure PAD in other versions of the same questionnaire (other languages), a cross-cultural adaptation and statistical validation of the questionnaire from English to Spanish will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* With a diagnosis of Peripheral Arterial Disease (intermittent claudication and critical lower limb ischemia)
* Whose first language is Spanish
* Who sign the informed consent.

Exclusion Criteria:

* Patients with cognitive impairment that difficults understanding of the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the Angiology and Vascular Surgery consultation
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Reliability | 3 -4 weeks from basal
  Reliability refers to the degree to which an instrument is capable of measuring without errors. It measures the proportion or variation in the measurements that is due to the diversity of values adopted by the variable and not to the possible systematic or random error. Reliability will be assessed trough Cronbach's alpha coefficient measured for every item of the questionnaire.
Reproducibility | 3-4 weeks from basal
  Reproducibility of intra-observer reliabilty refers to the repeatibility of the instrument, when it is administered with the same method to the same population at two times. Kappa Index will be measured
Validity | 3-4 weeks from basal
  Validity is the ability of the questionnaire to measure the construct for which it has been designed. Pearson correlation between the domains of the questionnaire and ABI from each patient will be measured

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Jimenez Diaz Foundation University Hospital, Madrid
  - La Paz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Olmedo JMD, Mendoza JAP, Reina-Bueno M. Revisión sistemática sobre el impacto de las complicaciones podológicas de la diabetes mellitus sobre la calidad de vida. Rev Esp Podol. 2017;28(1):30-6.
- [Background] Guyatt GH, Feeny DH, Patrick DL. Measuring health-related quality of life. Ann Intern Med. 1993 Apr 15;118(8):622-9. doi: 10.7326/0003-4819-118-8-199304150-00009. PMID 8452328
- [Background] Schwartzmann L. CALIDAD DE VIDA RELACIONADA CON LA SALUD: ASPECTOS CONCEPTUALES. Cienc Enferm. diciembre de 2003;9(2):09- 21.
- [Background] Guía de Consenso Multidisciplinar en Enfermedad Arterial Periférica de extremidades inferiores - Acta Sanitaria.
- [Background] Serrano Hernando FJ, Martin Conejero A. [Peripheral artery disease: pathophysiology, diagnosis and treatment]. Rev Esp Cardiol. 2007 Sep;60(9):969-82. doi: 10.1157/13109651. Spanish. PMID 17915154
- [Background] Soria-Juan B, Escacena N, Capilla-Gonzalez V, Aguilera Y, Llanos L, Tejedo JR, Bedoya FJ, Juan V, De la Cuesta A, Ruiz-Salmeron R, Andreu E, Grochowicz L, Prosper F, Sanchez-Guijo F, Lozano FS, Miralles M, Del Rio-Sola L, Castellanos G, Moraleda JM, Sackstein R, Garcia-Arranz M, Garcia-Olmo D, Martin F, Hmadcha A, Soria B; Collaborative Working Group "Noma Project Team". Cost-Effective, Safe, and Personalized Cell Therapy for Critical Limb Ischemia in Type 2 Diabetes Mellitus. Front Immunol. 2019 Jun 4;10:1151. doi: 10.3389/fimmu.2019.01151. eCollection 2019. PMID 31231366
- [Background] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901
- [Background] Morgan MB, Crayford T, Murrin B, Fraser SC. Developing the Vascular Quality of Life Questionnaire: a new disease-specific quality of life measure for use in lower limb ischemia. J Vasc Surg. 2001 Apr;33(4):679-87. doi: 10.1067/mva.2001.112326. PMID 11296317
- [Background] Poku E, Duncan R, Keetharuth A, Essat M, Phillips P, Woods HB, Palfreyman S, Jones G, Kaltenthaler E, Michaels J. Patient-reported outcome measures in patients with peripheral arterial disease: a systematic review of psychometric properties. Health Qual Life Outcomes. 2016 Nov 24;14(1):161. doi: 10.1186/s12955-016-0563-y. PMID 27881127
- [Background] Nordanstig J, Wann-Hansson C, Karlsson J, Lundstrom M, Pettersson M, Morgan MB. Vascular Quality of Life Questionnaire-6 facilitates health-related quality of life assessment in peripheral arterial disease. J Vasc Surg. 2014 Mar;59(3):700-7. doi: 10.1016/j.jvs.2013.08.099. Epub 2013 Dec 15. PMID 24342060
- [Background] de Almeida Correia M, Andrade-Lima A, Mesquita de Oliveira PL, Domiciano RM, Ribeiro Domingues WJ, Wolosker N, Puench-Leao P, Ritti-Dias RM, Cucato GG. Translation and Validation of the Brazilian-Portuguese Short Version of Vascular Quality of Life Questionnaire in Peripheral Artery Disease Patients with Intermittent Claudication Symptoms. Ann Vasc Surg. 2018 Aug;51:48-54.e1. doi: 10.1016/j.avsg.2018.02.026. Epub 2018 May 15. PMID 29772330
- [Background] Frans FA, van Wijngaarden SE, Met R, Koelemay MJ. Validation of the Dutch version of the VascuQol questionnaire and the Amsterdam Linear Disability Score in patients with intermittent claudication. Qual Life Res. 2012 Oct;21(8):1487-93. doi: 10.1007/s11136-011-0060-z. Epub 2011 Nov 15. PMID 22083223
- [Background] Ramada-Rodilla JM, Serra-Pujadas C, Delclos-Clanchet GL. [Cross-cultural adaptation and health questionnaires validation: revision and methodological recommendations]. Salud Publica Mex. 2013 Jan-Feb;55(1):57-66. doi: 10.1590/s0036-36342013000100009. Spanish. PMID 23370259
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN study reached international consensus on taxonomy, terminology, and definitions of measurement properties for health-related patient-reported outcomes. J Clin Epidemiol. 2010 Jul;63(7):737-45. doi: 10.1016/j.jclinepi.2010.02.006. PMID 20494804
- [Background] Aday LA, Cornelius LJ, Steven F, Cohen B, Aday LA, Cornelius LJ, et al. Published by Jossey-Bass.
- [Background] Carvajal A, Centeno C, Watson R, Martinez M, Rubiales AS. [How is an instrument for measuring health to be validated?]. An Sist Sanit Navar. 2011 Jan-Apr;34(1):63-72. doi: 10.4321/s1137-66272011000100007. Spanish. PMID 21532647
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Perneger TV, Courvoisier DS, Hudelson PM, Gayet-Ageron A. Sample size for pre-tests of questionnaires. Qual Life Res. 2015 Jan;24(1):147-51. doi: 10.1007/s11136-014-0752-2. Epub 2014 Jul 10. PMID 25008261
- [Background] Piault E, Doshi S, Brandt BA, Angun C, Evans CJ, Bergqvist A, Trocio J. Linguistic validation of translation of the Self-Assessment Goal Achievement (SAGA) questionnaire from English. Health Qual Life Outcomes. 2012 Apr 23;10:40. doi: 10.1186/1477-7525-10-40. PMID 22525050
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752